CLINICAL TRIAL: NCT04973488
Title: Therapeutic Plasma Exchange Followed by Convalescent Plasma Transfusion in Severe and Critically Ill COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novacescu Alexandru (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Sponsor-Investigator, Novacescu Alexandru, Director of trial - Supervisor, University of Medicine and Pharmacy "Victor Babes" Timisoara
Organization: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDYTPECVP20
Record Dates: First submitted 2021-07-20; First posted 2021-07-22 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection; Acute Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Therapeutic Plasma Exchange; Convalescent Plasma
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Single group, that is divided into two arms
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Not masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): In the treatment arm, Therapeutic plasma exchange will be conducted in the first 24 hours after being admitted into the intensive care unit, after which convalescent plasma from donors that have had COVID-19 will be transfused
  Interventions: Other: Therapeutic plasma exchange
- Control arm (No Intervention): In the control arm, patients will receive standard COVID-19 treatment

INTERVENTIONS:
Other: Therapeutic plasma exchange — The intervention is a combination between the procedure of Therapeutic plasma exchange and biological transfusion of convalescent plasma from donors that have have COVID-19
  Other Names: Transfusion of convalescent plasma
  Arms: Treatment arm

SUMMARY:
Therapeutic plasma exchange (TPE) has been proposed as a rescue therapy in critically ill COVID-19 patients. The aim of this study is to determine whether combining TPE with convalescent plasma (CVP) transfusion early during the intensive care unit (ICU) stay, improves survival among this heterogeneous population.

DETAILED DESCRIPTION:
This single centre prospective, non-randomised controlled trial will be conducted in an 8 bed COVID-19 ICU and will include patients with severe COVID-19 pneumonia requiring ICU monitoring and therapy. 19 patients will be treated performing TPE followed by CVP transfusion while for 19 patients will receive standard treatment according to hospital protocols. TPE will be initiated during the first 24 hours after ICU admission, followed immediately by transfusion of CVP. The primary endpoint is survival at 30 days. Secondary endpoints include assessing the evolution of biomarkers, such as the partial pressure of arterial oxygen (PaO2) to fractional inspired oxygen (FiO2) ratio (P/F ratio), C reactive protein (CRP), lactate dehydrogenase (LDH) and ferritin at the 7-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* positive reverse transcriptase PCR test for COVID 19
* COVID-19 pneumonia
* All patients included were adults (>18 years)
* Acute respiratory failure

Exclusion Criteria:

* pregnant women
* patients with suspected or confirmed pulmonary embolism
* patients with terminal disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Licker, MD, PhD, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (1):
- Municipal Hospital "Dr. Teodor Andrei" Lugoj, Lugoj, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Yes
We plan on sharing treatment protocol, demographic data of the study cohort, primary outcomes, secondary outcomes, miscellaneous data, treatment scheme, statystical data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available at 6 months after registering the study. It will be available for 36 months
Access Criteria: Data will be shared with interested researchers, contact: novacescu_alex@yahoo.com

REFERENCES:
- [Derived] Novacescu AN, Duma G, Buzzi B, Baditoiu LM, Bedreag O, Papurica M, Sandesc D, Sorescu T, Vlad D, Licker M. Therapeutic plasma exchange followed by convalescent plasma transfusion in severe and critically ill COVID-19 patients: A single centre non-randomized controlled trial. Exp Ther Med. 2022 Jan;23(1):76. doi: 10.3892/etm.2021.10999. Epub 2021 Nov 24. PMID 34934447
- See also: World Health Organization. WHO Coronavirus (COVID-19) Dashboard. Geneva: 2021 — https://covid19.who.int
- See also: Lin L, Li TS. [Interpretation of "Guidelines for the diagnosis and treatment of novel coronavirus (2019-nCoV) infection by the national health commission (Trial Version 5)" ]. Zhonghua Yi Xue Za Zhi. 2020;100(0):E001 — https://www.yiigle.com/LinkIn.do?linkin_type=DOI&DOI=10.3760%2Fcma.j.issn.0376-2491.2020.0001
- See also: Franchini M, Liumbruno GM. Convalescent plasma for the treatment of severe COVID-19. Biol Targets Ther. 2021;15:31-38 — https://www.dovepress.com/convalescent-plasma-for-the-treatment-of-severe-covid-19-peer-reviewed-fulltext-article-BTT
- See also: Keith P, Day M, Perkins L, Moyer L, Hewitt K, Wells A. A novel treatment approach to the novel coronavirus: an argument for the use of therapeutic plasma exchange for fulminant COVID-19. Crit Care. 2020;24(1):1-3 — https://ccforum.biomedcentral.com/articles/10.1186/s13054-020-2836-4
- See also: Gucyetmez B, Atalan HK, Sertdemir I, et al. Therapeutic plasma exchange in patients with COVID-19 pneumonia in intensive care unit: a retrospective study. Crit Care. 2020;24(1):1-4 — https://ccforum.biomedcentral.com/articles/10.1186/s13054-020-03215-8
- See also: Sarfraz A, Singh-Makkar S, Sarfraz Z, et al. Therapeutic plasma exchange and COVID-19: a rapid review. Clin Immunol Immunother. 2020;6(4):1-5 — https://www.heraldopenaccess.us/openaccess/therapeutic-plasma-exchange-and-covid-19-a-rapid-review
- See also: Kamran SM, Mirza ZE, Naseem A, et al. Therapeutic plasma exchange for coronavirus disease-2019 triggered cytokine release syndrome; a retrospective propensity matched control study. PLoS One. 2021;16(1 January):e0244853 — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0244853
- See also: Liu S, Lin H-M, Baine I, et al. Convalescent plasma treatment of severe COVID-19: a matched control study. Nat Med. 2020;26(11):1708-1713 — https://www.nature.com/articles/s41591-020-1088-9
- See also: Stahl K, Bode C, David S. First do no harm - beware the risk of therapeutic plasma exchange in severe COVID-19. Crit Care. 2020;24(1):1-2 — https://ccforum.biomedcentral.com/articles/10.1186/s13054-020-03070-7
- See also: Honore PM, Barreto Gutierrez L, Kugener L, et al. Plasma exchange in critically ill COVID-19 patients improved inflammation, microcirculatory clot formation, and hypotension, thereby improving clinical outcomes: Fact or fiction? Crit Care. 2020;24(1):1-2 — https://ccforum.biomedcentral.com/articles/10.1186/s13054-020-03262-1
- See also: Wang EY, Mao T, Klein J, et al. Diverse functional autoantibodies in patients with COVID-19. Nature. 2021;595:283-288 — https://www.nature.com/articles/s41586-021-03631-y
- See also: Fajnzylber J, Regan J, Coxen K, et al. SARS-CoV-2 viral load is associated with increased disease severity and mortality. Nat Commun. 2020;11(1):1-9 — https://www.nature.com/articles/s41467-020-19057-5

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients included in the study were adults (>18 years) who presented with acute respiratory failure and ARDS, had positive reverse transcriptase-polymerase chain reaction (RT-PCR) test results for SARS-CoV-2 virus and presented with clinical and/or radiological signs of COVID-19 pneumonia upon hospital admission. Exclusion criteria were represented by any of the following: Pregnancy, patients with suspected or confirmed pulmonary embolisms and patients with terminal disease.
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 7 | 21
  >=65 years | 5 | 12 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 19 | 19 | 38
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.75 (5.02) | 27.16 (6.92) | 28.45 (6.10)
Comorbidities present [Number; unit: participants] | 18 | 17 | 35
Symptoms onset to treatment [Mean (Standard Deviation); unit: Days] | 7.68 (2.49) | 8.58 (2.14) | 8.13 (2.33)
Acute Physiology and Chronic Health Evaluation (APACHE II) [Mean (Standard Deviation); unit: points] — The APACHE II score can be used to describe the morbidity of a patient when comparing the outcome with other patients.
  The APACHE II score ranges from 0 to 71 points. Increasing score is associated with increased mortality.
  points | 5.74 (3.16) | 7.58 (6.48) | 6.65 (5.11)
Severe form of COVID-19 [Count of Participants; unit: Participants] — The 'Guidelines for the Diagnosis and Treatment of Novel Coronavirus (2019-nCoV) Infection by the [Chinese] National Health Commission (Trial Version 5)' clinically distinguishes four levels of severity: Mild, common, severe and critical
  Participants | 12 | 10 | 22
Critical form of COVID-19 [Count of Participants; unit: Participants] — The 'Guidelines for the Diagnosis and Treatment of Novel Coronavirus (2019-nCoV) Infection by the [Chinese] National Health Commission (Trial Version 5)' clinically distinguishes four levels of severity: Mild, common, severe and critical
  Participants | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Number of Participants who Survived
Time Frame: 30 day period
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 19
Participants | 9 | 5

2. Secondary Outcome: P/F Ratio
Description: Average Partial pressure of arterial oxygen (PaO2) to fractional inspired oxygen (FiO2) ratio - P/F ratio calculated between the values from day 1 and day 7
Time Frame: 7 day period
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 19
ratio | 141.88 (37.19) | 109.61 (39.25)

3. Secondary Outcome: C Reactive Protein (CRP)
Description: Average value of CRP calculated using the values from day 1 and day 7
Time Frame: 7 day period
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 19
mg/l | 46.17 (60.89) | 144.00 (115.3)

4. Secondary Outcome: Lactate Dehydrogenase (LDH)
Description: Average value of LDH calculated using the values from day 1 and day 7
Time Frame: 7 day period
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 19
U/l | 375.11 (127.41) | 548.41 (218.03)

5. Secondary Outcome: Ferritin
Description: Average value of ferritin calculated using the values from day 1 and day 7
Time Frame: 7 day period
Measure: Mean (Standard Deviation); unit: micrograms/l
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 19
micrograms/l | 1563.23 (1206.05) | 1586.27 (1356.42)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Data regarding adverse event collection was obtained by the continuous monitoring of vital signs specific for the intensive care unit. During the treatment proposed in the intervention arm of this trial, a physician was supervising the vital signs of the patient to immediately stop the treatment in the event of an adverse event.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 10/19 | 14/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=19) | Control Arm (N=19)
Anaphylactic reaction (Cardiac disorders) | 1 (1) | 0 (0) — 1 patient in the treatment group presented with transient hypotension (systolic blood pressure <90 mmHg) after the transfusion of convalescent plasma, which resolved upon administration of crystalloid bolus.

LIMITATIONS AND CAVEATS:
Limitations of the study include the small number of patients enrolled and the non-randomized nature of the study. Also antibody titer was not determined in patients prior to the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT04973488/Prot_SAP_000.pdf